CLINICAL TRIAL: NCT00161187
Title: A Pilot Study of Irradiated HLA-Partially Matched Allogeneic Related Donor Lymphocytes for Patients With Selected Malignancies
Brief Title: Irradiated Donor Lymphocyte Infusion in Treating Patients With Relapsed or Refractory Hematologic Cancer or Solid Tumor
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Medicine and Dentistry of New Jersey (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: Rutgers, The State University of New Jersey (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 010101; P30CA072720 (NIH); 0220003330 (Other: CINJ IRB); CDR0000540298 (Other: NIH)
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2015-11-06 (Estimated); Status verified 2013-09

CONDITIONS: Cancer
Keywords: refractory chronic lymphocytic leukemia; recurrent small lymphocytic lymphoma; prolymphocytic leukemia; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; recurrent marginal zone lymphoma; splenic marginal zone lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; stage I multiple myeloma; stage II multiple myeloma; stage III multiple myeloma; recurrent mantle cell lymphoma; childhood diffuse large cell lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult Burkitt lymphoma; recurrent adult grade III lymphomatoid granulomatosis; recurrent childhood grade III lymphomatoid granulomatosis; adult nasal type extranodal NK/T-cell lymphoma; childhood nasal type extranodal NK/T-cell lymphoma; recurrent mycosis fungoides/Sezary syndrome; anaplastic large cell lymphoma; angioimmunoblastic T-cell lymphoma; recurrent adult T-cell leukemia/lymphoma; recurrent adult Hodgkin lymphoma; recurrent/refractory childhood Hodgkin lymphoma; recurrent adult acute myeloid leukemia; recurrent childhood acute myeloid leukemia; childhood chronic myelogenous leukemia; chronic phase chronic myelogenous leukemia; relapsing chronic myelogenous leukemia; recurrent renal cell cancer; stage IV renal cell cancer; recurrent bladder cancer; stage IV bladder cancer; recurrent prostate cancer; stage IV prostate cancer; recurrent malignant testicular germ cell tumor; stage III malignant testicular germ cell tumor; recurrent gastric cancer; stage IV gastric cancer; recurrent pancreatic cancer; stage IV pancreatic cancer; localized unresectable adult primary liver cancer; recurrent adult primary liver cancer; recurrent childhood liver cancer; recurrent colon cancer; stage IV colon cancer; recurrent rectal cancer; stage IV rectal cancer; recurrent breast cancer; stage IV breast cancer; extensive stage small cell lung cancer; recurrent non-small cell lung cancer; recurrent small cell lung cancer; stage IV non-small cell lung cancer; recurrent ovarian epithelial cancer; recurrent cervical cancer; recurrent adult soft tissue sarcoma; stage IV adult soft tissue sarcoma; chondrosarcoma; recurrent osteosarcoma; previously treated childhood rhabdomyosarcoma; recurrent childhood rhabdomyosarcoma; ovarian sarcoma; recurrent uterine sarcoma; stage IV uterine sarcoma; stage I small lymphocytic lymphoma; contiguous stage II small lymphocytic lymphoma; noncontiguous stage II small lymphocytic lymphoma; stage III small lymphocytic lymphoma; stage IV small lymphocytic lymphoma; accelerated phase chronic myelogenous leukemia; blastic phase chronic myelogenous leukemia; recurrent childhood large cell lymphoma; stage I childhood large cell lymphoma; stage II childhood large cell lymphoma; stage III childhood large cell lymphoma; stage IV childhood large cell lymphoma; adult primary hepatocellular carcinoma; advanced adult primary liver cancer; ovarian stromal cancer; stage IA cervical cancer; stage IB cervical cancer; stage IIA cervical cancer; stage IIB cervical cancer; stage III cervical cancer; stage IVA cervical cancer; stage IVB cervical cancer; recurrent adult acute lymphoblastic leukemia; untreated adult acute lymphoblastic leukemia; recurrent childhood acute lymphoblastic leukemia; untreated childhood acute lymphoblastic leukemia; recurrent endometrial carcinoma; stage I endometrial carcinoma; stage II endometrial carcinoma; stage III endometrial carcinoma; stage IV endometrial carcinoma; childhood hepatocellular carcinoma; stage III childhood liver cancer; stage IV childhood liver cancer; previously untreated childhood rhabdomyosarcoma; metastatic childhood soft tissue sarcoma; localized Ewing sarcoma/peripheral primitive neuroectodermal tumor; metastatic Ewing sarcoma/peripheral primitive neuroectodermal tumor; recurrent Ewing sarcoma/peripheral primitive neuroectodermal tumor; contiguous stage II grade 1 follicular lymphoma; contiguous stage II grade 2 follicular lymphoma; contiguous stage II grade 3 follicular lymphoma; noncontiguous stage II grade 1 follicular lymphoma; noncontiguous stage II grade 2 follicular lymphoma; noncontiguous stage II grade 3 follicular lymphoma; stage I grade 1 follicular lymphoma; stage I grade 2 follicular lymphoma; stage I grade 3 follicular lymphoma; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; contiguous stage II marginal zone lymphoma; noncontiguous stage II marginal zone lymphoma; stage I marginal zone lymphoma; stage III marginal zone lymphoma; stage IV marginal zone lymphoma; localized osteosarcoma; metastatic osteosarcoma; stage I ovarian epithelial cancer; stage II ovarian epithelial cancer; stage III ovarian epithelial cancer; stage IV ovarian epithelial cancer; recurrent ovarian germ cell tumor; stage I ovarian germ cell tumor; stage II ovarian germ cell tumor; stage III ovarian germ cell tumor; stage IV ovarian germ cell tumor; limited stage small cell lung cancer; refractory multiple myeloma; stage II malignant testicular germ cell tumor; stage I adult soft tissue sarcoma; stage II adult soft tissue sarcoma; stage III adult soft tissue sarcoma; stage I bladder cancer; stage II bladder cancer; stage III bladder cancer; male breast cancer; stage I breast cancer; stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer; stage I colon cancer; stage II colon cancer; stage III colon cancer; stage I gastric cancer; stage II gastric cancer; stage III gastric cancer; stage I non-small cell lung cancer; stage II non-small cell lung cancer; stage IIIA non-small cell lung cancer; stage IIIB non-small cell lung cancer; stage I pancreatic cancer; stage II pancreatic cancer; stage III pancreatic cancer; stage I prostate cancer; stage II prostate cancer; stage III prostate cancer; stage I rectal cancer; stage II rectal cancer; stage III rectal cancer; stage I renal cell cancer; stage II renal cell cancer; stage III renal cell cancer; stage I uterine sarcoma; stage II uterine sarcoma; stage III uterine sarcoma; stage I chronic lymphocytic leukemia; stage II chronic lymphocytic leukemia; stage III chronic lymphocytic leukemia; stage IV chronic lymphocytic leukemia; contiguous stage II mantle cell lymphoma; noncontiguous stage II mantle cell lymphoma; stage I mantle cell lymphoma; stage III mantle cell lymphoma; stage IV mantle cell lymphoma; Waldenstrom macroglobulinemia; contiguous stage II adult diffuse large cell lymphoma; noncontiguous stage II adult diffuse large cell lymphoma; stage I adult diffuse large cell lymphoma; stage III adult diffuse large cell lymphoma; stage IV adult diffuse large cell lymphoma; contiguous stage II adult Burkitt lymphoma; noncontiguous stage II adult Burkitt lymphoma; stage I adult Burkitt lymphoma; stage III adult Burkitt lymphoma; stage IV adult Burkitt lymphoma; stage I mycosis fungoides/Sezary syndrome; stage II mycosis fungoides/Sezary syndrome; stage III mycosis fungoides/Sezary syndrome; stage IV mycosis fungoides/Sezary syndrome; adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with t(15;17)(q22;q12); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with t(8;21)(q22;q22); untreated adult acute myeloid leukemia; untreated childhood acute myeloid leukemia and other myeloid malignancies; de novo myelodysplastic syndromes; secondary myelodysplastic syndromes; previously treated myelodysplastic syndromes; nonmetastatic childhood soft tissue sarcoma; recurrent childhood soft tissue sarcoma; stage I childhood Hodgkin lymphoma; stage II childhood Hodgkin lymphoma; stage III childhood Hodgkin lymphoma; stage IV childhood Hodgkin lymphoma; stage I adult Hodgkin lymphoma; stage II adult Hodgkin lymphoma; stage III adult Hodgkin lymphoma; stage IV adult Hodgkin lymphoma; recurrent childhood small noncleaved cell lymphoma; stage I childhood small noncleaved cell lymphoma; stage II childhood small noncleaved cell lymphoma; stage III childhood small noncleaved cell lymphoma; stage IV childhood small noncleaved cell lymphoma; Burkitt lymphoma; stage I adult T-cell leukemia/lymphoma; stage II adult T-cell leukemia/lymphoma; stage III adult T-cell leukemia/lymphoma; stage IV adult T-cell leukemia/lymphoma; stage I malignant testicular germ cell tumor; childhood myelodysplastic syndromes; childhood renal cell carcinoma; stage IA melanoma; stage IB melanoma; stage IIA melanoma; stage IIB melanoma; stage IIC melanoma; stage IIIA melanoma; stage IIIB melanoma; stage IIIC melanoma; stage IV melanoma; recurrent melanoma
MeSH Terms: conditions — Neoplasms; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Prolymphocytic; Lymphoma, B-Cell, Marginal Zone; Lymphoma, Follicular; Multiple Myeloma; Lymphoma, Mantle-Cell; Lymphoma, Large B-Cell, Diffuse; Burkitt Lymphoma; Lymphoma, Extranodal NK-T-Cell; Mycosis Fungoides; Sezary Syndrome; Lymphoma, Large-Cell, Anaplastic; Immunoblastic Lymphadenopathy; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Hodgkin Disease; Recurrence; Leukemia, Myeloid, Acute; Leukemia, Myeloid, Chronic-Phase; Carcinoma, Renal Cell; Urinary Bladder Neoplasms; Prostatic Neoplasms; Testicular Neoplasms; Stomach Neoplasms; Pancreatic Neoplasms; Carcinoma, Hepatocellular; Colonic Neoplasms; Rectal Neoplasms; Breast Neoplasms; Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma; Carcinoma, Ovarian Epithelial; Uterine Cervical Neoplasms; Sarcoma; Chondrosarcoma; Osteosarcoma; Leukemia, Myeloid, Accelerated Phase; Blast Crisis; Dendritic Cell Sarcoma, Interdigitating; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Endometrial Neoplasms; Neuroectodermal Tumors, Primitive, Peripheral; Breast Neoplasms, Male; Waldenstrom Macroglobulinemia; Congenital Abnormalities; Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (Experimental): Biological/Vaccine: therapeutic allogeneic lymphocytes The total CD3+ cell dose target is 1.8 x 108 CD3+ cells/kg +/- 1.0 x 108 CD3+ cells/kg. Up to 6 cycles.
  Interventions: Biological: therapeutic allogeneic lymphocytes

INTERVENTIONS:
Biological: therapeutic allogeneic lymphocytes — The total CD3+ cell dose target is 1.8 x 108 CD3+ cells/kg +/- 1.0 x 108 CD3+ cells/kg. Up to 6 cycles.

SUMMARY:
RATIONALE: When irradiated lymphocytes from a donor are infused into the patient they may help the patient's immune system kill cancer cells.

PURPOSE: This pilot study is looking at the side effects and how well irradiated donor lymphocyte infusion works in treating patients with relapsed or refractory hematologic cancer or solid tumor.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the toxicity of irradiated allogeneic donor lymphocyte infusion in patients with relapsed or refractory hematological cancer or solid tumor.
* Determine the response in patients treated with this regimen.
* Determine the presence of disease or antigen-specific lymphocytes in patients treated with this regimen.

OUTLINE: This is a pilot, open-label, controlled study.

Patients undergo irradiated allogeneic donor lymphocyte infusion over 1 hour on day 1. Treatment repeats every 8-16 weeks for up to 6 infusions in the absence of disease progression or unacceptable toxicity.

Blood samples are collected periodically and analyzed for lymphocytotoxicity directed towards patients' cells (normal and malignant cells) and for disease or antigen-specific cells. Samples are also analyzed for survival of donor lymphocytes by chimerism studies.

PROJECTED ACCRUAL: A total of 40 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed diagnosis of 1 of the following:

  * Hematologic cancer, including any of the following:

    * Chronic lymphocytic leukemia or small lymphocytic lymphoma meeting any of the following criteria:

      * Relapsed within 1 year after prior fludarabine phosphate-containing regimens OR not a candidate to receive such therapy due to comorbidities or allergies
      * Received prior anti-CD52 monoclonal antibody therapy OR ineligible to receive such therapy (for patients without symptomatic lymphadenopathy)
      * Has documentation of disease-associated symptoms, rapid progression of disease, or other indications for treatment
    * B- or T-cell prolymphocytic leukemia meeting any of the following criteria:

      * Relapsed within 1 year after prior fludarabine phosphate- or alkylating agent-containing regimens OR not a candidate to receive such therapy due to comorbidities or allergies
      * Relapsed within 1 year after prior anti-CD20 monoclonal antibody therapy OR ineligible to receive such therapy (for patients with CD20-positive disease)
      * Received prior anti-CD52 monoclonal antibody therapy OR ineligible to receive such therapy (for patients without symptomatic lymphadenopathy)
    * Lymphoplasmacytic lymphoma, marginal zone lymphoma, mucosa-associated lymphoid tissue lymphoma, or follicular lymphoma meeting any of the following criteria:

      * Relapsed within 1 year after prior fludarabine phosphate- or alkylating agent-containing regimens or radioconjugated anti-CD20 monoclonal antibody OR not a candidate to receive such therapy due to comorbidities or allergies
      * Relapsed within 1 year after prior anti-CD20 monoclonal antibody therapy OR ineligible to receive such therapy (for patients with CD20-positive disease)
      * Has documentation of disease-associated symptoms, rapid progression of disease, or other indications for treatment
    * Multiple myeloma meeting any of the following criteria:

      * Relapsed after prior alkylating agents, thalidomide, corticosteroids, or bortezomib OR not a candidate to receive such therapy due to comorbidities or allergies
      * Relapsed after prior high-dose chemotherapy followed by autologous hematopoietic stem cell rescue OR not a candidate to receive such therapy
    * Mantle cell lymphoma that has relapsed after prior combination chemotherapy or anti-CD20 monoclonal antibody OR not a candidate to receive such therapy
    * Diffuse large B-cell lymphoma meeting any of the following criteria:

      * Relapsed after prior salvage combination chemotherapy with or without high-dose chemotherapy followed by autologous hematopoietic stem cell rescue OR not a candidate to receive such therapy
      * Received prior radiolabeled anti-CD20 monoclonal antibody OR ineligible to receive such therapy (for patients with transformed large cell lymphoma)
    * Burkitt's lymphoma

      * Relapsed after prior salvage combination chemotherapy with or without high-dose chemotherapy followed by autologous hematopoietic stem cell rescue OR not a candidate for such therapy
    * Lymphomatoid granulomatosis or mature T-cell or NK-cell neoplasms meeting any of the following criteria:

      * Relapsed after prior single agent or combination chemotherapy OR not a candidate to receive such therapy
      * Has documentation of disease-associated symptoms, rapid progression of disease, or other indications for treatment
    * Mycosis fungoides or Sezary syndrome

      * Relapsed after prior combination chemotherapy, interferon-α, denileukin diftitox, or extracorporeal photophoresis OR not a candidate to receive such therapy
    * Anaplastic large cell lymphoma, peripheral T-cell lymphoma unspecified, or angioimmunoblastic T-cell lymphoma meeting the following criteria:

      * Relapsed after prior salvage combination chemotherapy with or without high-dose chemotherapy followed by autologous hematopoietic stem cell rescue OR not a candidate to receive such therapy
    * Hepatosplenic T-cell lymphoma or adult T-cell leukemia/lymphoma

      * Relapsed after prior salvage combination chemotherapy OR not a candidate to receive such therapy
    * Hodgkin's lymphoma

      * Relapsed after prior salvage combination chemotherapy with or without high-dose chemotherapy followed by autologous hematopoietic stem cell rescue OR not a candidate to receive such therapy
    * Acute lymphocytic leukemia meeting any of the following criteria:

      * Relapsed during or after prior multi-agent combination chemotherapy administered in sequential induction, consolidation, and maintenance courses OR not a candidate to receive such therapy
      * Relapsed after prior salvage combination chemotherapy with or without high-dose chemotherapy followed by autologous hematopoietic stem cell rescue OR not a candidate to receive such therapy
      * Relapsed after prior chemotherapy with or without radiotherapy followed by allogeneic hematopoietic stem cell transplant (or ineligible for such therapy) AND demonstrates persistent cytogenetic, fluorescent in situ hybridization (FISH), or molecular (reverse transcriptase-polymerase chain reaction) evidence of bcr-abl fusion gene despite 6 weeks of treatment with imatinib mesylate
    * Acute myelogenous leukemia or myelodysplasia meeting any of the following criteria:

      * Relapsed or refractory disease after prior induction chemotherapy (anthracycline and cytarabine, topotecan hydrochloride and cytarabine, or comparable regimen) OR not a candidate to receive such therapy
      * Not a candidate for chemotherapy with or without radiotherapy followed by allogeneic or autologous hematopoietic stem cell transplant
      * Patients with acute promyelomonocytic leukemia must have received prior tretinoin and arsenic trioxide
    * Chronic myelogenous leukemia meeting any of the following criteria:

      * Relapsed or refractory disease after prior imatinib mesylate
      * Not a candidate for chemotherapy with or without radiotherapy followed by allogeneic hematopoietic stem cell transplant
      * Chronic phase disease allowed if there is FISH or cytogenetic evidence of increasing disease
  * Solid tumor, including any of the following:

    * Renal cell carcinoma

      * Metastatic relapsed or refractory disease after prior high-dose aldesleukin OR ineligible to receive such therapy due to comorbidities OR did not consent to treatment
    * Bladder cancer or gastric cancer

      * Metastatic relapsed or refractory disease after prior combination therapy OR not a candidate to receive such therapy
    * Prostate cancer

      * Metastatic relapsed or refractory disease after prior hormonal therapy OR not a candidate to receive such therapy
    * Testicular cancer

      * Metastatic relapsed or refractory disease after prior standard induction or salvage chemotherapy or high-dose chemotherapy with autologous hematopoietic stem cell rescue OR not a candidate to receive such therapy
    * Pancreatic cancer

      * Metastatic relapsed or refractory disease after prior gemcitabine hydrochloride-based therapy OR not a candidate to receive such therapy
    * Hepatocellular carcinoma

      * Unresectable or metastatic disease
    * Colorectal carcinoma

      * Metastatic relapsed or refractory disease after prior combination therapy, including fluorouracil with or without leucovorin calcium, oxaliplatin, or irinotecan hydrochloride OR not a candidate to receive such therapy
    * Breast cancer meeting any of the following criteria:

      * Metastatic relapsed or refractory disease after prior first- or second-line standard combination chemotherapy OR not a candidate to receive such therapy
      * Received prior trastuzumab (Herceptin®) and sequential hormonal therapy OR not a candidate to receive such therapy as indicated by the biological characteristics of the cancer
    * Lung cancer (non-small cell or small cell lung cancer), ovarian cancer, endometrial cancer, or cervical cancer

      * Metastatic relapsed or refractory disease after prior first- or second-line combination chemotherapy OR not a candidate to receive such therapy
    * Malignant melanoma

      * Metastatic relapsed or refractory disease after prior immunotherapy or combination chemotherapy OR not a candidate to receive such therapy
    * Sarcoma meeting any of the following criteria:

      * Metastatic relapsed or refractory disease after prior first- or second-line combination chemotherapy OR not a candidate to receive such therapy
      * Not a candidate for resection
      * Patients with gastrointestinal stromal tumors must have received prior imatinib mesylate
* Measurable disease
* Must have received prior available standard therapy for specific disease OR not a candidate for this treatment
* No CNS malignancy
* HLA-partially matched (≥ 2/6 HLA antigen [A, B, DR]) related donor (above 18 years of age) available

PATIENT CHARACTERISTICS:

* ECOG performance status 0-1
* Life expectancy > 3 months
* Bilirubin < 1.5 times upper limit of normal (ULN)
* AST < 3.0 times ULN
* LVEF > 35%
* No active infections
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No uncontrolled medical or psychiatric illness that would preclude study compliance, in the opinion of the investigator

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2001-05; Primary Completion 2010-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Toxicity | 10 years

SECONDARY OUTCOMES:
Response | 10 years
Presence of disease or antigen-specific lymphocytes | 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Roger Strair, MD, PhD, Principal Investigator — Rutgers Cancer Institute of New Jersey
Locations (1):
- Cancer Institute of New Jersey at UMDNJ - Robert Wood Johnson Medical School, New Brunswick, New Jersey, United States